CLINICAL TRIAL: NCT04712123
Title: Recurrent S. Aureus Infections in Osteoarticular Infections
Acronym: RELAPSTAPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 281
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Staphylococcus Aureus Infection; Bone and Joint Infection
Keywords: Staphylococcus Aureus Infection; Bone and Joint Infection; relapse
MeSH Terms: conditions — Staphylococcal Infections; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- relapse due to S. aureus: patients having had an initial infection due to S. aureus and who present a relapse with persistence of S. aureus
  Interventions: Other: relapse due to S. aureus

INTERVENTIONS:
Other: relapse due to S. aureus — to find out if it is the same S. aureus in both infections

SUMMARY:
Staphylococcus aureus osteoarticular infections, in particular those associated with the presence of implant, relapse in 20% of cases. Currently, the reasons for these relapses are poorly understood, whether on the microbiological or clinical side.

The aim of this study is to improve knowledge on persistence of mechanisms of S. aureus

ELIGIBILITY:
Inclusion Criteria:

* patients having had an osteoarticular infection with or without material due to S. aureus presenting a recurrence of S. aureus infection

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients having had an osteoarticular infection with or without material due to S. aureus and treated at CRIOAc Lyon, presenting a recurrence of S. aureus infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of patients having had an osteoarticular infection due to S. aureus | between 2015 and 2020
  proportion of patients having had an osteoarticular infection due to S. aureus
Description of patients having had an osteoarticular infection due to S. aureus | between 2015 and 2020
  type of patients: age, BMI, comorbidities...
Description of Bone and Joint Iinfection/Prosthesis Joint Infection | between 2015 and 2020
  implant or prosthesis or not, acute/ chronic, bacteriology

SECONDARY OUTCOMES:
rate of patients having had a relapse due to persistence of S. aureus | between 2015 and 2020
  proportion of patients having had an osteoarticular infection due persistence of S. aureus
rate of S. aureus strain identical between the initial episode and the relapse | between 2015 and 2020
  proportion of relapse due to the same strain of S. aureus than in the initial episode

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/